CLINICAL TRIAL: NCT05199909
Title: Prospective, Single Arm and Open Clinical Observation of Zanubrutinib in the Treatment of Antiphospholipid Syndrome With Secondary Thrombocytopenia
Brief Title: Safety and Efficacy of Zanubrutinib in the Treatment of Antiphospholipid Syndrome With Secondary Thrombocytopenia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2021048
Record Dates: First submitted 2021-12-30; First posted 2022-01-20 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-01

CONDITIONS: Antiphospholipid Syndrome; Thrombocytopenia; Treatment
MeSH Terms: conditions — Antiphospholipid Syndrome; Thrombocytopenia | interventions — zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intervention ( zanubrutinib) (Experimental): 10 enrolled patients are picked up to take zanubrutinib at the indicated dose.
  Interventions: Drug: zanubrutinib

INTERVENTIONS:
Drug: zanubrutinib — The initial dose is 80mg/day. If the treatment is ineffective after 4 weeks, and under the condition of good safety, the researcher will judge that the dosage should be added to 80mg twice/day，or a higher dose for oral maintenance. The maximum dose is 160mg twice a day. The duration of zanubrutinib is 24 weeks.
  In case of intolerable adverse reactions, such as severe infection, severe bleeding, hematopenia, arrhythmia, etc., investigator can reduce the dose of zanubrutinib, or withdraw from clinical trials as appropriate.
  Other Names: The treatment of zanubrutinib

SUMMARY:
To evaluate the safety and efficacy of zanubrutinib in the treatment of antiphospholipid syndrome with secondary thrombocytopenia in 10 patients.

DETAILED DESCRIPTION:
Antiphospholipid syndrome (APS) is a disease spectrum characterized by thrombosis and/or pathological pregnancy, and characterized by persistent antiphospholipid antibodies (APL) positive in laboratory examination. The incidence of thrombocytopenia in APS patients is 29.6%. Thrombocytopenia is usually mild to moderate without clinical manifestations, and the risk of bleeding is low. The platelet count of most patients is > 50 × 10^9/L. If APS has severe thrombocytopenia and severe bleeding, it is very difficult to treat it. According to previous literature reports, Some patients were treated with hormones, rituximab and immunosuppressants. Platelets can be obviously increased, but they are easy to relapse and difficult to maintain. aPL is not obviously decreased and difficult to be completely eliminated. Thrombosis still occurs in some patients with obviously decreased platelets. Thrombopoietin receptor agonists increase the risk of thrombosis, which is a difficult point in hematology treatment at present.

Bruton tyrosine kinase (BTK), a member of the Tec family of non-receptor tyrosine kinases, is expressed in all hematopoietic cells except T cells and terminal differentiated plasma cells. BTK is a key kinase in BCR signaling pathway, which regulates B cell proliferation, survival, differentiation and cytokine expression. BTK inhibitors can affect autoimmune diseases (AID) involving B cells and non-B cells through B cell receptor, Fc receptor and RANK receptor signals, such as systemic lupus erythematosus (SLE), multiple sclerosis (MS) and rheumatoid arthritis (RA).

Besides its activity in B cells, BTK is also expressed in platelets and mediates the signal of cell surface receptor glycoprotein VI (GPVI). It is believed that BTK/Tec pathway may affect GP VI specific platelet signal deficiency and interfere with collagen adhesion and vWF-mediated platelet activation. BTK plays an important role in vWF-mediated signal transduction and GPIb-dependent thrombosis in vivo. Moreover, recent studies have found that BTK inhibitors can block the activation of platelets stimulated by FcγRIIA through antibody-mediated crosslinking (inducing platelet aggregation and secretion) or anti-CD9 antibody (only inducing platelet aggregation). Therefore, BTK inhibitors have certain antithrombotic effects at the same time. At present, there is no related report on BTK inhibitor in the treatment of APS abroad. BTK inhibitors can regulate B cell proliferation, survival, differentiation and cytokine expression, reduce antibody formation, and inhibit platelet adhesion and platelet activation, so they may have a good therapeutic effect on antiphospholipid syndrome.

Therefore, the investigators designed this clinical trial to provide a new treatment option for the clinical treatment of antiphospholipid syndrome with secondary thrombocytopenia.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above, male or female；
* Diagnosis of antiphospholipid syndrome；
* Failure to receive glucocorticoid treatment in the past (the curative effect cannot be maintained, or recurs, or cannot be tolerated); Can not choose other second-line treatment, such as rituximab, cyclosporine, cyclophosphamide, etc.; Or rituximab, cyclosporine and other treatments are ineffective, relapsed or intolerable;
* Plt < 30×10^9/L；
* Liver and kidney function, such as ALT, AST, BUN, SCR < 1.5 × upper limit of normal value, passing physical examination;
* ECOG physical state score ≤ 2 points；
* Cardiac function of the New York Society of Cardiac Function ≤ 2；
* Signed and dated written informed consent.

Exclusion Criteria:

* Uncontrollable primary diseases of important organs, such as malignant tumors, liver failure, heart failure, renal failure and other diseases；
* HIV positive;
* Accompanied by uncontrollable active infection, including hepatitis B, hepatitis C, cytomegalovirus, EB virus and syphilis positive;
* Accompanied by extensive and severe bleeding, such as hemoptysis, upper gastrointestinal hemorrhage, intracranial hemorrhage, etc.;
* At present, there are heart diseases, arrhythmias that need treatment or hypertension that researchers judge is poorly controlled;
* Patients with thrombotic diseases such as new pulmonary embolism and unstable period of various arteriovenous thrombosis;
* Those who have received allogeneic stem cell transplantation or organ transplantation in the past;
* Patients with mental disorders who cannot normally obtain informed consent and conduct trials and follow-up;
* Patients whose toxic symptoms caused by pre-trial treatment have not disappeared;
* Other serious diseases that may limit the subject's participation in this test (such as diabetes; Severe cardiac insufficiency; Myocardial obstruction or unstable arrhythmia or unstable angina pectoris in recent 6 months; Gastric ulcer，etc.);
* Patients with septicemia or other irregular severe bleeding;
* Pregnant women, suspected pregnancies (positive pregnancy test for human chorionic gonadotropin in urine at screening) and lactating patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-01-25 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with a platelet count ≥ 30 × 10^9/L and 50×10^9/L at week 12(Day 85) | 12 weeks
  Observe the changes of blood routine platelet count after 12 weeks of treatment, and calculate the proportion and times of subjects ≥ 30 × 10^9/L and 50 × 10^9/L.

SECONDARY OUTCOMES:
Persistent platelet response with clinical significance at 24 weeks | 24 weeks
  Response defined as as the proportion of subjects with platelet count ≥ 50 × 109/L in at least 4 of the last 6 visits within 24 weeks without rescue treatment.
Number of participants with clinically significant bleeding as assessed using the world health organization (WHO) bleeding scale. | 24 weeks
  The WHO Bleeding Scale is a measure of bleeding severity with the following grades: grade 0 = no bleeding, grade 1= petechiae, grade 2= mild blood loss, grade 3 = gross blood loss, and grade 4 = debilitating blood loss.
The occurrence of adverse events during treatment (AE/SAE), treatment-related adverse events (TRAE) and serious adverse events (TRSAE) | 24 weeks
  The occurrence of adverse events during treatment (AE/SAE), treatment-related adverse events (TRAE) and serious adverse events (TRSAE)
Evaluate the occurrence of thrombosis during treatment | 24 weeks
  Evaluate the occurrence of thrombosis during treatment
Antiphospholipid antibody titre | 24 weeks
  To monitor antiphospholipid antibody titre during treatment in all participants.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, MD, Principal Investigator — Chinese Academy of Medical Science and Blood Disease Hospital
Locations (2):
- China (2):
  - Chinese Academy of Medical Science and Blood Disease Hospital, Tianjin, Tianjin Municipality
  - Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Yes
Researchers qualified can request the dataset, including de-identified individual subject data. Data may be requested from PI from 12 months 36 months after study completion.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 months to 36 months after study completion.
Access Criteria: Upon request to PI.